CLINICAL TRIAL: NCT03882424
Title: A Randomized, Double-blind, Single-dose, Three-arm, Parallel-group, Phase 1 Study to Compare Pharmacokinetic and Safety of TRS003 to China-approved Bevacizumab and US-licensed Avastin®，When Administered to Healthy Male Participants
Brief Title: A Study to Compare Pharmacokinetic and Safety of TRS003 to China-approved Bevacizumab and US-licensed Avastin®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TRS00301001
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TRS003 (Experimental): Proposed biosimilar of bevacizumab，Intravenous administration
  Interventions: Biological: TRS003
- China-approved Bevacizumab (Active Comparator): Intravenous administration
  Interventions: Biological: China-approved Bevacizumab
- US-licensed Avastin (Active Comparator): Intravenous administration
  Interventions: Biological: US-licensed Avastin

INTERVENTIONS:
Biological: TRS003 — 25mg/mL (4 mL/vial) Injection，Single dose of 3mg/kg Intravenous infusion for 90 minutes
  Arms: TRS003
Biological: China-approved Bevacizumab — 25mg/mL (4 mL/vial) Injection，Single dose of 3mg/kg Intravenous infusion for 90 minutes
  Arms: China-approved Bevacizumab
Biological: US-licensed Avastin — 25mg/mL (4 mL/vial) Injection，Single dose of 3mg/kg Intravenous infusion for 90 minutes
  Arms: US-licensed Avastin

SUMMARY:
This is a 12-week, randomized, double-blind, single-dose pharmacokinetic (PK) study. Approximately 114 healthy male participants (screening occurred within 28 days prior to dosing) will be randomized 1:1:1 to either TRS003, China-approved bevacizumab, and US-licensed Avastin® groups. Study drug will be dispensed as a single 3 mg/kg dose for intravenous infusion within 90 minutes. PK and immunogenicity samples will be collected and safety will be assessed. The primary objective of this study was to demonstrate pharmacokinetic similarity between TRS003, China-approved bevacizumab and US-licensed Avastin®, as measured by AUC0-inf in healthy male participants after a single 3 mg/kg dose.

DETAILED DESCRIPTION:
The primary assessment of PK similarity will be based upon a 90 percentage confidence interval (CI) for the ratio of the geometric means (TRS003, China-approved bevacizumab and US-licensed Avastin®) for AUC0-inf on PK analysis set. If the 90 percentage CI of the ratio of the geometric means for AUC0-inf is within the range of 80-125 percentage, then PK similarity will be concluded. Secondary PK parameters such as but not limited to Cmax, AUClast will be analyzed using the same statistical approach. A nonparametric approach, for example, Wilcoxon signed-rank test, will be taken to evaluate parameters such as t1/2. Exploratory analyses may be performed for other PK parameters as deemed appropriate. All adverse events (AEs) will be listed and summarized using descriptive methodology. The incidence of AEs for each treatment will be presented by severity and association with the study drugs. Clinical laboratory parameters, vital signs, and electrocardiogram (ECG) parameters will be listed and summarized using descriptive statistics. The number and percentage of participants testing positive for anti-drug antibodies (ADAs) will be summarized by treatment and time point.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male participants, 18-55 years old with no significant medical history, and in good health as determined by detailed medical history, full physical examination, vital signs, 12-lead electrocardiogram (ECG), urinalysis and laboratory tests at screening.
* Body mass index of 17.5-30.5 kg/m^2 and body weight of 50-95 kg.
* Protocol-specified hematology, coagulation, blood chemistry and urinalysis within the laboratory normal range at screening, unless deemed not clinically significant by the Investigator.
* Participants must have adequate organ function according to the following laboratory values:

  1. Bone marrow function (absolute neutrophil count ≥1500/mm^3 and platelet count ≥100,000/mm^3)
  2. Adequate liver function [alanine aminotransferase (ALT) ≤3 × upper limit normal (ULN) and alkaline phosphatase ≤2 × ULN, total bilirubin ≤1.5 mg/dL]
  3. Adequate renal function creatinine clearance ≥60 mL/min based on Cockcroft-Gault equation
* Participants must agree to use an acceptable form of birth control throughout the study and for at least 18 weeks after the study is over.

Exclusion Criteria:

* Participants unable to give voluntary informed consent.
* Evidence or history of clinically significant disease, cancer other than adequately treated basal cell or squamous cell carcinoma of the skin.
* Participants on anticoagulant drugs, anemic or with known bleeding diatheses.
* Participants with a history of severe, uncontrolled hypertension, heart disease, cerebrovascular incidents, gastrointestinal bleeding, hemoptysis, frequent epistaxis or gingival bleeding.
* History clinically significant orthostatic hypotension, fainting spells, vasovagal syncope.
* Uncontrolled severe hypertension (140/90 mm Hg).
* Previous treatment with an anti-VEGF antibody or any other antibody or protein targeting the VEGF receptor.
* Use of any prescription, investigational drugs, herbal supplements or nonprescription drugs within 1 month or 5 half-lives (whichever is longer) prior to the first dose, or dietary supplements within 1 week prior to the first dose. If needed, paracetamol/acetaminophen may be used, but must be documented in the Concomitant medications/Significant non-drug therapies page of the case report form (CRF).
* Serious unhealed wound, cutaneous ulcer or bone fracture at the time of screening.
* Major surgery or major dental procedure or significant traumatic injury within 2 months prior to screening, or any planned surgery or procedure within 3 months after investigational treatment administration. Participants must have recovered from all acute surgery- or trauma-related complications.
* Participant's medical and family history of recent or recurrent thromboembolism or other clotting and coagulation disorders.
* Donated blood over 400 mL within 3 months.
* History of relevant and clinically significant intra-abdominal inflammation, gastrointestinal perforation or gall bladder perforation.
* History of severe allergic or anaphylactic reaction to a therapeutic drug or severe seasonal allergies.
* Recent (within the last three [3] years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* A positive hepatitis B, hepatitis C or HIV tests at screening indicative of a current or past infection.
* Current use of tobacco or nicotine-containing products. Concomitant treatment was given only if Investigator believes strictly necessary and should be documented.
* Current use of any biologic drugs.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 114 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smith Robina, MD, Principal Investigator — WCCT Global, Inc.
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Started | 38 | 38 | 38
Completed | 34 | 38 | 38
Not Completed | 4 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — schedule conflict | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin | Total
Number analyzed (Participants) | 38 | 38 | 38 | 114
Age, Customized [Count of Participants; unit: Participants]
  Safety Population: <18 | 0 | 0 | 0 | 0
  Safety Population: 18-40 | 26 | 30 | 25 | 81
  Safety Population: >40 | 12 | 8 | 13 | 33
  Pharmacokinetic Population: <18 | 0 | 0 | 0 | 0
  Pharmacokinetic Population: 18-40 | 26 | 30 | 25 | 81
  Pharmacokinetic Population: >40 | 12 | 8 | 13 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 38 | 38 | 38 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 27 | 25 | 79
  Not Hispanic or Latino | 11 | 11 | 13 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 15 | 22 | 25 | 62
  Race: Black | 18 | 8 | 9 | 35
  Race: Asian | 4 | 6 | 4 | 14
  Race: Am Indian | 1 | 0 | 0 | 1
  Race: Hawaiian | 0 | 0 | 0 | 0
  Race: Multi-racial | 0 | 0 | 0 | 0
  Race: Other | 0 | 2 | 0 | 2
Height [Mean (Full Range); unit: cm] | 175.37 [163.0 to 188.2] | 173.09 [161.3 to 181.5] | 174.62 [155.4 to 184.6] | 174.36 [155.4 to 188.2]
Weight [Mean (Full Range); unit: kg] | 80.16 [62.6 to 92.8] | 78.55 [57.1 to 94.5] | 78.82 [59.7 to 94.7] | 79.18 [57.1 to 94.7]
BMI [Mean (Full Range); unit: kg/m^2] | 26.09 [20.6 to 30.4] | 26.21 [20.4 to 30.5] | 25.84 [20.0 to 30.5] | 26.05 [20.0 to 30.5]

OUTCOME MEASURES:

1. Primary Outcome: AUC0-inf，Area Under the Serum Concentration Versus Time Curve，Time 0 to Infinity
Description: The primary assessment of PK similarity will be based upon a 90 percentage CI for the ratio of the geometric means (TRS003, China-approved bevacizumab and US-licensed Avastin®) for AUC0-inf on PK analysis set. If the 90 percentage CI of the ratio of the geometric means for AUC0-inf is within the range of 80-125 percentage, then PK similarity will be concluded.
Time Frame: Pre-dose, 0 hour (End of infusion, EOI), 0.5 hour, 4 hours, 8 hours, 24 hours, 48 hours, 96 hours, 168 hours, 336 hours, 672 hours, 1008 hours, 1344 hours, 1680 hours, and 2016 hours post EOI
Measure: Geometric Least Squares Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Number analyzed (Participants) | 34 | 38 | 38
hr*ng/mL | 30308695.01 (4780171.58) | 28449241.04 (5232124.54) | 29050169.73 (4476342.82)

2. Secondary Outcome: Cmax, Maximum Drug Concentration
Description: To assess other PK parameters such as Cmax, following a single dose of TRS003, China-approved bevacizumab and US-licensed Avastin® in healthy male participants. If the 90 percentage CI of the ratio of the geometric means for Cmax is within the range of 80-125 percentage, then PK similarity will be concluded.
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Number analyzed (Participants) | 38 | 38 | 38
ng/mL | 86051.02 (14888.99) | 84748.14 (12592.56) | 82509.03 (13197.95)

3. Secondary Outcome: AUC0-last, Area Under the Serum Concentration-time Curve，Time 0 to Last
Description: To assess other PK parameters such as AUClast, following a single dose of TRS003, China-approved bevacizumab and US-licensed Avastin® in healthy male participants. If the 90 percentage CI of the ratio of the geometric means for AUC0-last is within the range of 80-125 percentage, then PK similarity will be concluded.
Time Frame: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Number analyzed (Participants) | 34 | 38 | 38
hr*ng/mL | 29146948.37 (4383124.30) | 27446018.92 (4716128.56) | 27951588.98 (4089884.99)

4. Secondary Outcome: Number of Participants Who Develop Detectable Anti-drug Antibody (ADA)
Description: To determine the number of participants with immunogenicity against TRS003, China-approved bevacizumab, and US-licensed Avastin® in healthy male participants, blood samples will be collected for ADA analyses.
Time Frame: Pre-dose, 336 hours, 672 hours, 1344 hours and 2016 hours after EOI (End of infusion)
Population: In TRS003, four subjects were lost to follow-up and one subject elected to withdraw due to schedule conflict, resulting in 13 samples missing.
  In China-approved bevacizumab, three subjects were lost to follow-up, resulting in 4 samples missing.
  In US-licensed Avastin, two subjects were lost to follow-up, resulting in 2 sample missing.
Measure: Count of Participants; unit: Participants
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Number analyzed (Participants) | 38 | 38 | 38
Participants
  0 hour: Negative | 37 | 37 | 38
  0 hour: Positive | 1 | 1 | 0
  336 hour: number analyzed (Participants) | 36 | 37 | 37
  336 hour: Negative | 36 | 37 | 37
  336 hour: Positive | 0 | 0 | 0
  672 hour: number analyzed (Participants) | 35 | 37 | 37
  672 hour: Negative | 35 | 37 | 37
  672 hour: Positive | 0 | 0 | 0
  1344 hour: number analyzed (Participants) | 33 | 36 | 38
  1344 hour: Negative | 33 | 34 | 38
  1344 hour: Positive | 0 | 2 | 0
  2016 hour: number analyzed (Participants) | 35 | 38 | 38
  2016 hour: Negative | 35 | 35 | 38
  2016 hour: Positive | 0 | 3 | 0

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse events will be classified using the MedDRA classification system. The severity of the toxicities will be graded according to the NCI CTCAE version 4.03.
Time Frame: Within 85 days following the drug administration
Population: 110 subjects completed the study. Three subjects who received Treatment A (Subject Nos. Subject Nos. 1-119, 1-120, and 1-177) were lost to follow-up and 1 subject (Subject No. 1-138) who received Treatment A was withdrawn from the study due to other reason (schedule conflict).
Measure: Count of Participants; unit: Participants
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
Number analyzed (Participants) | 38 | 38 | 38
Participants | 6 | 12 | 11

ADVERSE EVENTS:
Time Frame: Throughout the study, subjects were monitored for AEs. All AEs, including those reported within 85 days following the last dose of drug administration, were recorded. AEs were followed-up until complete resolution, or until the Medical Sub-Investigator judged safe to discontinue follow-up. Any subjects who were withdrawn from the study due to an AE were followed until the outcome of the AE was determined.
Arm/Group | TRS003 | China-approved Bevacizumab | US-licensed Avastin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 6/38 | 12/38 | 11/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRS003 (N=38) | China-approved Bevacizumab (N=38) | US-licensed Avastin (N=38)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03882424/Prot_003.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03882424/SAP_004.pdf